CLINICAL TRIAL: NCT02201511
Title: A Phase 1, Open-label Study In Healthy Subjects To Investigate the Pharmacokinetics Of Pf-06412562 Following Single Oral Administration Of Modified Release Formulation In Fasted And Fed States
Brief Title: A Healthy Volunteer Trial to Gain Information About the Blood Concentrations of PF-06412562 After Oral Administration of a Modified Release Formulation in Fasted and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7441006; 2014-001214-25 (EudraCT Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: relative bioavailbility; food effect; pharmacokinetics; ALTERATION OF COGNITIVE FUNCTIONS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: 3 mg PF-06412562 MR tablets_Fasted
- 2 (Experimental)
  Interventions: Drug: 2 x 15 mg PF-06412562 MR tablets_Fasted
- 3 (Experimental)
  Interventions: Drug: 2 x 15 mg PF-06412562 MR tablets_Fed
- 4 (Experimental)
  Interventions: Drug: 10 mg PF-06412562 IR tablets

INTERVENTIONS:
Drug: 3 mg PF-06412562 MR tablets_Fasted — A single modified release tablet with 3 mg PF-06412562 administered after an overnight fast
  Arms: Arm 1
Drug: 2 x 15 mg PF-06412562 MR tablets_Fasted — Two 15 mg PF-06412562 modified release tablets administered after an overnight fast
  Arms: 2
Drug: 2 x 15 mg PF-06412562 MR tablets_Fed — Two 15 mg PF-06412562 modified release tablets administered after a high fat breakfast
  Arms: 3
Drug: 10 mg PF-06412562 IR tablets — a single immediate release tablet of 10 mg PF-06412562 after an overnight fast
  Arms: 4

SUMMARY:
The study is designed to understand the blood concetration of PF-06412562 and its metabolite, PF-06663872, following a single oral dose of a modified release formulation. The study will include two doses of the PF-06412562 modified release formulation to understand the proportionality. Effect of food on absorption of PF-06412562 from the modified release formulation will also be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs);

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* Subjects who have attempted suicide in the past.
* Subjects who have an unexplained history of sudden death in their family

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0-2 days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-2 days
Time after dose and before the first plasma concentration (Tlag) | 0-2
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf] | 0- 2 days
  AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. It is obtained from AUC (0 - t) plus AUC (t - inf).
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 0-2 days
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Plasma Decay Half-Life (t1/2) | 0-2 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441006&StudyName=A%20healthy%20volunteer%20trial%20to%20gain%20information%20about%20the%20blood%20concentrations%20of%20PF-06412562%20after%20oral%20administration%20of%20a%20modified%20rele